CLINICAL TRIAL: NCT03442140
Title: Harmonica Playing Improves Inspiratory and Expiratory Muscle Strength, Reduces Shortness of Breath With Activity, and Improves Quality of Life in Patients With COPD
Brief Title: Harmonica Playing Improves Quality of Life in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 017-135
Record Dates: First submitted 2018-02-08; First posted 2018-02-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: COPD
Keywords: COPD; Shortness of breath; Harmonica
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients who completed the Baylor Martha Foster Lung Center Pulmonary Rehabilitation Program at least six months ago will participate in the 12-week harmonica program
  Interventions: Other: Harmonica playing

INTERVENTIONS:
Other: Harmonica playing — Patients will play the harmonica for up to 6 months

SUMMARY:
15 patients who have completed the Baylor Martha Foster Lung Center Pulmonary Rehabilitation Program at least six months ago will be selected to participate in a 12 week training program with six months of follow up.

DETAILED DESCRIPTION:
Subjects will be consented and evaluated prior to beginning the Harmonica Training. Subjects will undergo spirometry testing, six minute walk testing and inspiratory capacity, inspiratory and expiratory respiratory muscle strength will be measured. A music therapist will evaluate their ability to assess the participant's ability to play the harmonica and offer assistance during the training. Subjects will complete a self-reported depression, shortness of breath, and quality of life questionnaire. All evaluations and questionnaires will be completed before and after the 12 week program and six months after the training program.

They will be trained to play the Harmonica and practice as a group during a twelve week program, for one hour a day, one day a week with the Instructors, one is a Registered Respiratory Therapist and the other is a music therapist, who will evaluate their ability and offer assistance. The music therapist will meet individually with each study participant at the beginning of the study to assess participants' harmonica playing ability.

They are required to practice at home (individually) in between classes for 30 minutes five days a week outside the formal training hour with the group. They may use oxygen as prescribed by their physician during the training. The training booklet includes information to help the subject with COPD understand how this program is designed to help them. They will also be given instructions on how to clean the harmonica and infection control measures to use during the program to prevent infections that could occur using the harmonica.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to attend 12 weeks of harmonica training for one hour a day per week
* Practice playing at home 30 minutes x 5 days a week
* Documented diagnosis of COPD
* Ability to perform spirometry, IC, MIP, and MEP maneuver and 6 minute walk
* Willing to complete depression, quality of life, shortness of breath, functional evaluation questionnaires
* Willing to perform in a group setting

Exclusion Criteria:

* Current COPD exacerbation
* Inability to perform spirometry, IC, MIP and MEP maneuver
* Inability to commit to weekly one hour sessions for 12 weeks and practice for 5 days/week.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Reduction in Shortness of Breath | 6 months
  Change 6-minute walk test and spirometry from baseline to 12 weeks and 6 months.

SECONDARY OUTCOMES:
saint George Quality of Life | 6 months
  Change in self-reported measures on St. George quality of life questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Millard, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States